CLINICAL TRIAL: NCT06176118
Title: Clinical Trial of 2-HOBA in Pulmonary Arterial Hypertension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, James D. West, Professor-Allergy, Pulmonary, and Critical Care Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230458
Record Dates: First submitted 2023-11-30; First posted 2023-12-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: 2-hoba; Pulmonary Hypertension; Right Ventricular
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Unblinded Intervention (Experimental): There is no control group in this study. Only intervention group due to phase of trial and study intentions.
  Interventions: Dietary Supplement: 2-HOBA

INTERVENTIONS:
Dietary Supplement: 2-HOBA — 2-HOBA supplement take three times daily for 12-weeks

SUMMARY:
Based on existing literature and clinical trials, 2- hydroxbenzylamine (2-HOBA) has clear impact on mechanisms that much of the international field of pulmonary hypertension (PH) research agrees are central to disease progression. The investigator's preliminary data and Phase I studies demonstrate not only a clear positive impact on reducing pulmonary vascular resistances in Group I and II PH, and both cytokine and molecular biomarkers of disease, but also indicated the potential for a substantial positive effect on heart function under load stress. In this Phase II project, investigators will test the safety and efficacy of 2-HOBA in PH patients, improving the function of the right ventricle under stress in a large animal model, and effectiveness in the context of standard-of-care in mouse models and large animals, to establish the remaining data needed to proceed to commercialization.

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH) is a disease in which gradual cellular occlusion of the blood vessels in the lungs increases pulmonary vascular resistance, eventually leading to right heart failure and death. Approved therapies in common use are all different classes of vasodilator, which can extend life in some patients, but are not disease modifying and do not prevent decline and death. There is thus need for new therapies for PH.

Although originating causes are different across patients, a common molecular factor across most etiologies is an increase in reactive oxygen species leading to a set of specific metabolic problems. These include increased insulin resistance, increased reliance on glutamine uptake in the lungs, a shift away from normal TCA-glucose metabolism, and suppressed fatty acid oxidation in the heart leading to increased intracellular fat. An important part of the mechanism is a feedback loop in which ROS causes reactive lipids particularly within the mitochondria, which then adduct to proteins causing loss of function and further metabolic defects. One such target in PH is the mitochondrial lysine deacetylase, Sirt3. In a recent clinical trial attempting an intervention on this metabolic axis, the only patients in whom it succeeded were those with an unusual activating set of SNPs in Sirt3, indicating that rescue of Sirt3 is a prerequisite for resolving disease.

This presents the possibility of rescuing the defects in metabolic function that are required for disease progression by alleviating the upstream problem with reactive lipid species. 2-Hydroxybenzylamine (2-HOBA) is a potent scavenger of reactive lipid dicarbonyls. It blocks the effects of reactive lipids by selectively trapping them - giving an alternate target to bind to with a binding affinity two to three orders of magnitude stronger. We have published that 2-HOBA treatment rescued Sirt3 activity in vivo in BMPR2 mutant mice, resulting in normalization of metabolic markers and near normalization of pulmonary vascular resistance2, resulting in reduced acetylation of key targets. In Phase I of this project, we found that 2-HOBA also reduced pulmonary pressures in the AKR-high fat diet model of Group II PH, the most common form of disease, associated with metabolic syndrome. The investigators also identified cytokines and metabolites known to be changed in PH that were corrected in our models, which could be used as biomarkers. Metabolic changes in the hearts in response to 2-HOBA in both mouse models which the investigators believe are extremely positive - increased ability to metabolize fatty acids, which is a key need in the right ventricle under stress.

The investigator's preliminary studies show that 2-HOBA is a safe compound which shows great promise in treating the core molecular defect in PH, in both the closest genetic mouse model to human disease available (BMPR2 mutants), in a mouse model of the most common type of PH (AKR-high fat diet) and in existing and animal toxicity and human safety trials.

Based on existing literature and clinical trials, 2- hydroxbenzylamine (2-HOBA) has clear impact on mechanisms that much of the international field of pulmonary hypertension (PH) research agrees are central to disease progression. Our preliminary data and Phase I studies demonstrate not only clear positive impact on reducing pulmonary vascular resistances in Group I and II PH, and both cytokine and molecular biomarkers of disease, but also indicated the potential for a substantial positive effect on heart function under load stress. In this Phase II project, investigators will test the safety and efficacy of 2-HOBA in PH patients, improving function of the right ventricle under stress in a large animal model, and effectiveness in the context of standard-of-care in mouse models and large animals, to establish the remaining data needed to proceed to commercialization.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older
* Diagnosed with idiopathic, heritable, simple congenital heart defect, or drug- or toxin-associated pulmonary arterial hypertension (PAH) according to World Health Organization consensus recommendations.
* Stable PAH-specific medication regimen for three months prior to enrollment. Subjects with only a single diuretic adjustment in the prior three months will be included. Adjustments in IV prostacyclin for side effect management are allowed.
* FEV1> or = 60% predicted and no more than mild abnormalities on lung imaging
* WHO Functional Class II-IV
* Ambulatory

Exclusion Criteria:

* Sensitivity to 2-HOBA
* Sensitivity to aspirin or salicylates
* Aspirin-related rhinitis or wheezing
* Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting angina, activity-limiting osteoarthritis, or other condition that limits activity
* Pregnancy
* Diagnosis of PAH etiology other than idiopathic, heritable, simple congenital heart defect, or associated with drugs or toxins
* Drug and toxin associated PAH patients with active drug use
* Prior diagnosis of cirrhosis
* Malignancy
* eGFR by MDRD <60mL/min
* Non-english speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in acetylated SOD2 and LCAD in plasma | baseline and 12-weeks
  This is a direct indication of effect; the mechanism of action of 2-HOBA is sequestration of lipids, and so this will demonstrate that it is having the desired molecular effect.

SECONDARY OUTCOMES:
Change in plasma LDL, HDL, triglyceride, free fatty acid concentration measured as a concentration (mg/dL) | baseline and 12-weeks
  Plasma concentrations based measures in mg/dL
Change in plasma acylcarnitine profile measured as a concentration (mg/dL) | baseline and 12-weeks
Change in meters walked in six-minute walk distance (meters) | baseline and 12-weeks
  The 6MWT measures the distance (in meters), a participant can walk at a comfortable speed on a flat, hard surface in 6 minutes. The intent of the 6MWD test is to evaluate exercise capacity associated with carrying out daily physical activities.
Change in Quality of Life as measured by the emPHasis-10 | baseline and 12-weeks
  The emPHasis-10 is a short and easy questionnaire that consists of 10 items that address breathlessness, fatigue, control, and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Change in Estimated Right Ventricle (RV) Systolic Pressure, as assessed by echocardiogram results, expressed in mmHg | baseline and 12-weeks
Change in Right Ventricle (RV) Free Wall Longitudinal Strain, as assessed by echocardiogram results, and expressed as percent (%) change in myocardial deformation. | baseline and 12-weeks
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | baseline and 12-weeks